CLINICAL TRIAL: NCT03642730
Title: Interactive Guided Ultrasound Examinations Done by Non-experts of Ultrasound Imaging
Acronym: EPISODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ICBE-2-11984
Record Dates: First submitted 2018-05-09; First posted 2018-08-22 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Disease; Heart Failure; Cardiac Ischemia
Keywords: echocardiography; training; follow-up
MeSH Terms: conditions — Heart Diseases; Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Masking Description: Masking is not applicable, since software study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scanned patients (Experimental): Scanned patients TransThoracic Echocardiography Diagnostic Test: TransThoracic Echocardiography imaging synchronized with additional external sensors
  Interventions: Device: TransThoracic Echocardiography imaging
- Non-expert scanning volunteers (Experimental): Non-expert scanning volunteers (among the medical staff at the clinical site) TransThoracic Echocardiography Diagnostic Test: TransThoracic Echocardiography imaging synchronized with additional external sensors
  Interventions: Device: TransThoracic Echocardiography imaging

INTERVENTIONS:
Device: TransThoracic Echocardiography imaging — ultrasound scanning

SUMMARY:
This prospective study is a pilot study for evaluating a guidance system that aims to facilitate high-quality echocardiographic acquisitions.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the feasibility for non-expert users (medical professionals but non-certified sonographers) to acquire parasternal, apical and subcostal views of suitable quality by using an existing ultrasound device (CE-marked, available in the market) and an additional guidance system (software prototype + probe motion tracking device). Such a system will help the user to place the probe on the patient and provide guidance for optimal acquisition of parasternal, apical and subcostal views.

The secondary objective of this study is to assess the feasibility for non-expert users to reproduce a simple clinical protocol by using an existing ultrasound device and the same additional guidance system.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers must have the ability to provide informed consent.
* All volunteers should be affiliated to the French Social Security.
* All volunteers will be scheduled for a routine transthoracic echocardiography exam in the echocardiography laboratory at the investigation site as part of standard care.

Exclusion Criteria:

* Subjects with congenital heart diseases (except bicuspid aortic valve)
* Pregnant women
* Adults lacking decisional capacity
* Adults placed under a legal protection regime (guardianship, curatorship, judicial protection)
* Adults not affiliated to the French Social Security
* Adults in emergent or critical condition
* Adults with active pain in the intended scanning region
* Adults with active skin disease or lesions in the intended scanning region
* Adults with allergy/sensitivity to ultrasound gel

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Echocardiography acquisition score [in %] [Operator's outcome] | Day 1
  Composite measurement that characterizes the echocardiography acquisition of the operator who is being assessed with respect to a 2D reference acquisition The echocardiography acquisition score is a combination of the view type score and the image quality score
Time to acquisition [in seconds] [Operator's performance] | Day 1
  Time to acquisition [in seconds] to reach an echocardiography acquisition score of 25%, 50%, 75% and 90%
Displacement [in mm] of the echocardiography probe with respect to the 2D reference acquisition [Technical reproducibility] | Day 1
  Displacement [in mm] of the echocardiography probe at the acquisition time with respect to the 2D reference acquisition [Reproducibility of the probe position and orientation]
Displacement [in mm] of the echocardiography probe with respect to the ideal acquisition [Geometrical reliability] | Day 1
  Displacement [in mm] of the echocardiography probe at the acquisition time with respect to the ideal (geometrical) acquisition estimated from 3D reference acquisition [Geometrical reliability of the probe position and orientation]

SECONDARY OUTCOMES:
Left ventricular Ejection Fraction [in %] [Measurement reproducibility] | Day 1
  Left ventricular Ejection Fraction [in %] by Simpson's biplane method

CONTACTS AND LOCATIONS:
Overall Officials: Eric Saloux, MD, Principal Investigator — Hospital
Locations (1):
- CHU Caen Service de Cardiologie, Caen, France

IPD SHARING:
Plan to Share IPD: No